CLINICAL TRIAL: NCT04705558
Title: Combination of Ketogenic Diet and Aerobic Exercise Versus Ketogenic Diet Alone in Prediabetes Female With Normal Weight
Brief Title: Combination of Ketogenic Diet and Exercise on Prediabetes in Female With Normal Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Abdelkhalek, lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KETO , EXERCISE ON PREDIABETES
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: two intervention:combination of continuous aerobic exercise in form of treadmill 5 sessions per week and ketogenic diet.
  ketogenic diet alone.
Who Masked: Participant, Investigator
Masking Description: double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): Continuous aerobic exercise with ketogenic diet for three month
  Interventions: Other: continuous moderate intensity aerobic training; Other: ketogenic diet
- group II (Experimental): Ketogenic diet alone for three month
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Other: continuous moderate intensity aerobic training — continuous moderate intensity aerobic exercises with ketogenic diet group underwent supervised moderate-intensity exercised on a treadmill at 50%-70% of heart rate reserve for three month
  Arms: group I
Other: ketogenic diet — Ketogenic diet: a low carbohydrate high-fat diet consisted of the following nutrient conformation: 80% fat, 15% protein and 5% carbohydrates, entire daily intake was estimated to be 20-30 g of carbohydrates for three month.

SUMMARY:
Individuals with prediabetes have a high risk of developing type 2 diabetes. The purpose of this study was to compare the effect of combination of ketogenic diet and aerobic exercise interventions versus ketogenic diet alone on the glucose level in prediabetes female with normal weight.

DETAILED DESCRIPTION:
Pre-diabetes is the preceding condition of diabetes, where the blood sugar level is higher than normal but lower than the diagnostic criteria of type II diabetes and in most of the cases, this ultimately leads to the development type II diabetes. It has been estimated that the number of pre-diabetic cases will increase to more than 470 million people worldwide, and this is understandably a worrying trend . Many studies have been done on diabetes patients. However, little is known about the pre-diabetic conditions.

Diagnosed Prediabetes was stated as any participants who did not have diabetes but who had fasting plasma glucose level of 100 - 125 mg/dL, an HbA1c level of 5.7% - 6.4%, or 2-hour plasma glucose level of 140 - 199 mg/dL.

Treatment of pre-diabetes and prevention of the development of pre-diabetes to T2DM,through lifestyle intervention mainly includes nutritious dietary and exercises.

Combining a ketogenic diet with exercise is a powerful way to reducing insulin resistance, control blood glucose levels and achieve weight loss. As ketogenic diets are nowadays predictable as being useful, there is presently a shortage of research studies examining just how useful the combination of exercise and a ketogenic diet

ELIGIBILITY:
Inclusion criteria:

1. female with their age ranged from 40-60 years
2. body mass index (BMI) from 20-25 kg/m2
3. fasting serum glucose range 5.6 to 6.9 mmol/L
4. hemoglobin A1C value fell within the prediabetes range (5.7%-6.4%) without medications, or treatment with oral hypoglycemic agents and/or insulin.

Exclusion criteria:

1. renal insufficiency
2. liver disease
3. abnormal cardiovascular function
4. diabetes
5. untreated hypertension
6. dyslipidemia
7. abnormal thyroid function
8. anyone who has undergone gallbladder removal
9. musculoskeletal constraint preventing them from fully participating in the exercise intervention

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female with prediabetes
Enrollment: 70 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-02-07 (Estimated); Study Completion 2021-02-10 (Estimated)

PRIMARY OUTCOMES:
change in fasting plasma glucose | three month
  Fasting blood specimen was obtained and measured participants' fasting plasma glucose.
  Diagnosed Prediabetes was stated as any participants who did not have diabetes but who had fasting plasma glucose level of 5.6 - 7.0 mmol/L
change in glycated hemoglobin | three month
  Fasting blood specimen was obtained and measured participants' glycated hemoglobin (HbA1c) Diagnosed Prediabetes was stated as any participants who did not have diabetes but who had HbA1c level of 5.7% - 6.4%

SECONDARY OUTCOMES:
change in Body composition | three month
  Body Weight was measured in kilograms and Height was measured in meters then body mass index (BMI) was calculated by dividing weight in kilograms on height in meters square BMI = kg/m2 .
  Waist circumference measurements have been made to the nearest 0.1 centimeter using a tape measure at the uppermost lateral border of the hip crest (ilium)

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Abdelkhalek, Cairo, Egypt